CLINICAL TRIAL: NCT00706771
Title: A Randomized Double-blind Controlled Pilot Feasibility and Safety Trial of NGAL-directed Sodium Bicarbonate to Protect Renal Function in Patients With the Systemic Inflammatory Response Syndrome, Oliguria and Elevated Lipocalin Levels
Brief Title: Bicarbonate and Lipocalin in Systemic Inflammatory Response Syndrome (SIRS) Study
Acronym: BLISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of Intensive Care Research, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNH 18/08
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Oliguria; Renal Impairment
Keywords: sodium bicarbonate; serum neutrophil gelatinase associated lipocalin; renal impairment; renal failure; systemic inflammatory response syndrome; defined; by serum NGAL ≥ 100 ng/ml.
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Oliguria; Renal Insufficiency | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium bicarbonate (Active Comparator): sodium bicarbonate: loading of 0.5 mmol/kg and the continuous infusion o f0.2 mmol/kg/hr
  Interventions: Drug: Sodium bicarbonate
- Sodium chloride (Active Comparator): sodium chloride: loading of 0.5 mmol/kg and the continuous infusion o f0.2 mmol/kg/hr
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate: loading dose of 0.5 mmol/Kg and then continuous infusion of 0.2 mmol/Kg/hr
  Arms: Sodium bicarbonate
Drug: Sodium chloride — 0.9% sodium chloride: loading dose of 0.5 mmol/Kg and then continuous infusion of 0.2 mmol/Kg/hr
  Arms: Sodium chloride

SUMMARY:
The investigators will determine the feasibility, safety and efficacy of intravenous sodium bicarbonate in reducing progression to overt acute renal failure in patients with the systemic inflammatory response syndrome, and low urine output or early acute renal impairment as defined by serum neutrophil gelatinase-associated lipocalin (NGAL).

DETAILED DESCRIPTION:
The investigators hypothesise:

1. In patients with SIRS and oliguria the early administration of sodium bicarbonate or sodium chloride (control) triggered by an abnormally high NGAL level is feasible.
2. In patients with SIRS and oliguria the early administration of sodium bicarbonate or sodium chloride (control) triggered by an abnormally high NGAL level is safe.
3. In patients with SIRS and oliguria the early administration of sodium bicarbonate or sodium chloride (control) triggered by an abnormally high NGAL level leads to signs or trends of efficacy as measured by serum creatinine derived indices.

ELIGIBILITY:
Inclusion Criteria:

* Consent obtained
* Diagnosis of SIRS. Requires any TWO of:

temperature > 38°C or < 36°C OR heart rate > 90 beats/min OR respiratory rate > 20 breaths/min. PaCO2 < 32 mm Hg OR alteration of white blood cell count > 12,000 cells/mm3, < 4,000 cells/mm3, or the presence of > 10% immature neutrophils

* elevated lipocalin level
* Arterial line already in place
* Central venous catheter already in place
* Age ≥ 18 years
* Within 24 hours of admission to the ICU

Exclusion Criteria:

* Unlikely to remain in ICU for >72 hours
* Moribund patient
* Pre-existing CKD, transplant or ESRD
* Receiving (or about to receive) continuous renal replacement therapy for acute renal failure at time of enrolment
* Diagnosis of acute GN, AIN, vasculitis or post-renal aetiology
* Known/suspected study allergy to sodium bicarbonate
* Enrolling physician concern about patient enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The ability to deliver the study protocol safely and rapidly with a trend to improved renal outcomes | 28 days

SECONDARY OUTCOMES:
Attenuation in lipocalin levels | 28 days
Decrease in the magnitude in serum creatinine rise | 28 days
Ability to deliver the study protocol without significant biochemical side effects | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Reade, MBBS DPhil, Principal Investigator — Austin & Northern Hospitals, University of Melbourne; Nerina Harley, MBBS FCICM, Principal Investigator — Melbourne Health; Rinaldo Bellomo, MD FJFICM, Principal Investigator — Austin Hospital, University of Melbourne
Locations (2):
- Australia (2):
  - Austin Hospital, Heidelberg, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria